CLINICAL TRIAL: NCT00758550
Title: Visual Function After Bilateral Implantation of AcrySof® Toric
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Benny Li, Scientific Clinical Affairs Manager, Alcon Research Ltd.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CM-06-17
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Results first posted 2010-03-16 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2010-03

CONDITIONS: Visual Function
Keywords: Visual function;; Refractive cylinder;; AcrySof® Toric;; AcrySof® Natural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AcrySof Toric IOL (Experimental): AcrySof Toric Intraocular Lens (IOL)
  Interventions: Device: AcrySof® Toric IOL
- AcrySof Natural IOL (Active Comparator): AcrySof Natural Intraocular Lens (IOL)
  Interventions: Device: AcrySof Natural

INTERVENTIONS:
Device: AcrySof® Toric IOL — AcrySof® Toric Intraocular Lens (IOL) implanted into the study eye following cataract extraction surgery
  Arms: AcrySof Toric IOL
Device: AcrySof Natural — AcrySof Natural Intraocular Lens (IOL) implanted into the study eye following cataract extraction surgery
  Arms: AcrySof Natural IOL

SUMMARY:
The objective of this study was to evaluate visual function of AcrySof Toric and AcrySof Natural Intraocular Lenses (IOLs) following implant for replacement of cataract.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral cataracts
* 40~80 years of age
* 4 Days - 1 Week interval between a single patient's surgery
* dilated pupil size (in dim light) ≥ 4.0 mm
* Anticipated correction with an IOL of +10 Diopters ~ +25 Diopters
* 0.75 - 2.0 Diopters of astigmatism preoperatively as measured by Keratometry readings

Exclusion Criteria:

* Preoperative ocular pathology
* Previous intraocular or corneal surgery
* An increased risk for complications which could require vitreoretinal surgery
* Corneal irregularities
* Corneal opacities
* Current contact lens usage(within 6 months prior to first surgery)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-04; Primary Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 60 cataract patients were enrolled into the study
Pre-assignment Details: Randomized
Groups:
- AcrySof Toric IOL: AcrySof Toric Intraocular Lens
- AcrySof Natural IOL: AcrySof Natural Intraocular Lens
Period: Overall Study
Arm/Group | AcrySof Toric IOL | AcrySof Natural IOL
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AcrySof Toric IOL | AcrySof Natural IOL | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 15 | 27
  >=65 years | 18 | 15 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Uncorrected Visual Acuity (UCVA)
Description: Uncorrected Visual Acuity (UCVA) from surgery measured in logMAR. LogMAR is the "logarithm of the minimum angle of resolution". A lower logMAR value indicates better visual acuity.
Time Frame: 6 Months after surgery
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | AcrySof Toric IOL | AcrySof Natural IOL
Number analyzed (Participants) | 30 | 30
logMAR | 0.06 (0.14) | 0.14 (0.11)

2. Secondary Outcome: Questionnaire Results
Description: Results of questionnaire rating the quality of distance vision without glasses or contact lenses. Measured on a scale of 0 to 6 (0 = worst, 6 = best).
Time Frame: 6 Months
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | AcrySof Toric IOL | AcrySof Natural IOL
Number analyzed (Participants) | 30 | 30
Units on a scale | 5.6 (0.7) | 4.5 (0.7)

ADVERSE EVENTS:
Arm/Group | AcrySof Toric IOL | AcrySof Natural IOL
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No